CLINICAL TRIAL: NCT01442961
Title: Postoperative Pain After Vaginal or Laparoscopic Hysterectomy: a Prospective Trial
Brief Title: Vaginal Hysterectomy, Laparoscopic Hysterectomy, Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Arvi Yli-Hankala, professor, Tampere University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R09003
Record Dates: First submitted 2011-09-19; First posted 2011-09-29 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Postoperative Pain
Keywords: pain, postoperative; hysterectomy, vaginal; surgery, gynecological
MeSH Terms: conditions — Pain, Postoperative | interventions — Laparoscopy; Hysterectomy, Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- laparoscopy (Active Comparator): Intervention: Procedure: laparoscopy
  Interventions: Procedure: laparoscopy, laparoscopic hysterectomy
- vaginal (Active Comparator): Intervention: Procedure: vaginal
  Interventions: Procedure: vaginal : vaginal hysterectomy

INTERVENTIONS:
Procedure: laparoscopy, laparoscopic hysterectomy — laparoscopic hysterectomy
  Arms: laparoscopy
Procedure: vaginal : vaginal hysterectomy — Vaginal hysterectomy
  Arms: vaginal

SUMMARY:
The previous studies have shown that recovery after laparoscopic or vaginal hysterectomy is faster than after abdominal approach. The aim of this study is to evaluate postoperative pain after vaginal or laparoscopic hysterectomy. The primary outcome measurement is opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -69 years
* Gender . female
* ASA status 1-3
* Vaginal hysterectomy or laparoscopic hysterectomy

Exclusion Criteria:

* Body mass Index over 35
* Diabetes Mellitus
* Liver disease
* Allergies to pharmaceuticals used in the Study
* Present use of opioids
* Vaginal prolapse

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative consumption of an opioid (oxycodone) | 20 hours
  the consumption of oxycodone will be monitored by recording the amount of the drug received via a commercially available patient controlled analgesia (PCA) pump

SECONDARY OUTCOMES:
NRS (numeral rating scale) of pain | 20 hours
  NRS is evaluated frequently during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland